CLINICAL TRIAL: NCT03191279
Title: Førstehjelp Gjort av Lekfolk-effekt på dødelighet og behandlingsforløp (First Aid by Laypersons - Effect on Mortality and Length of Stay)
Brief Title: First Aid by Laypersons - Effect on Mortality and Length of Stay
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Tromso (Other)
Collaborators: University Hospital of North Norway (Other); Norsk Folkehjelp (Unknown); Nasjonal kompetansetjeneste for traumatologi (NKT-Traume) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2016/1760
Record Dates: First submitted 2017-05-03; First posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Wounds and Injury; First Aid; Bystander; Trauma
Keywords: Wounds and injury; Trauma; First aid; Bystander; Laypersons
MeSH Terms: conditions — Wounds and Injuries | interventions — First Aid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- First aid correct: Patient has received first aid according to local guidelines for all indicated first aid measures from bystanders on scene of accident when the first ambulance arrives
  Interventions: Procedure: First aid
- First aid attempted: Bystanders have attempted first aid for indicated first aid measures, but measures have been incorrectly performed according to local guidelines
  Interventions: Procedure: First aid
- No first aid: Indicated first aid measures have not been carried out when the first ambulance arrives on scene

INTERVENTIONS:
Procedure: First aid — Open airway (head tilt, chin lift), recovery position, staunch of bleeding, prevention of hypothermia, cooling of burn, CPR
  Groups: First aid attempted; First aid correct

SUMMARY:
The study aims to assess the effect of first aid from bystanders on survival, admission length, and need of ICU-stay for trauma victims.

DETAILED DESCRIPTION:
All ambulance services in Norway will be invited to participate. In the participating ambulance services, the personnel of first unit to reach the scene of accident for any emergency response to trauma will register what first aid measures (if any) are indicated and have been performed by the bystanders on the scene up til the point where the ambulance arrives. Hospital data for each case will be retrieved. Those patients who did receive correct first aid will then be compared to those patients who did not receive first aid, and those where first aid was attempted but not correct for differences in share of survivors, length of hospital stay, and need for admission to ICU.

ELIGIBILITY:
Inclusion Criteria:

* All emergency response calls to trauma (drownings and hangings included)

Exclusion Criteria:

* No injury to patient
* Non-traumatic condition
* Poisonings

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who has sustained an injury and where the EMS has been alerted and initiated an emergency response
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Admission length | 3 months after inclusion
  Length of hospital stay after injury, in days
Survival | 1 month after inclusion
  30-day survival, starting from day of injury
Need of ICU stay | 3 months after inclusion
  Whether patient is admitted to ICU during admission

SECONDARY OUTCOMES:
Length of ICU stay | 3 months after inclusion
  Length of ICU stay if patient was admitted to ICU, in days

OTHER OUTCOMES:
Whether patients received first aid from bystanders | At time of inclusion
  If patients with indicated measures receiving first aid from bystanders, given for each measure and combined
Whether first aid measures were indicated for the patient | At time of inclusion
  If first aid measures was indicated, given for each measure and combined

CONTACTS AND LOCATIONS:
Locations (1):
- UNN Tromsø, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No
No plan of sharing IDP